CLINICAL TRIAL: NCT00185575
Title: Duloxetine for the Treatment of Dysthymia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Lorrin M Koran, Principal Investigator, Stanford University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUSPO30478
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2009-04-09 (Estimated); Status verified 2009-04

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: duloxetine

SUMMARY:
The purpose of this study is to test the hypothesis that duloxetine (Cymbalta), in doses of 60 or 120 mg/day, is an effective and tolerable treatment for adult outpatients suffering from dysthymia. Dysthymia is chronic, mild depression characterized by feeling sad or low more days than not for more than 2 years.

DETAILED DESCRIPTION:
The purpose of this research is to obtain information on the safety and effectiveness of duloxetine (Cymbalta) in the treatment of dysthymia. Duloxetine has been approved by the federal Food and Drug Administration for the treatment of depression. The use of duloxetine for treatment of dysthymia is considered experimental.

Dysthymia is defined as chronic, low-grade depression, characterized by feeling low or depressed, that lasts for two or more years. Additional symptoms may include: poor appetite or overeating; insomnia or sleeping too much; low energy or fatigue; low self-esteem; poor concentration or difficulty making decisions; and feelings of hopelessness.

Dysthymia affects 3-6% of the general population, but is an underdiagnosed and undertreated disorder. In double-blind, placebo-controlled clinical trials of antidepressant medications, dysthymia response rates are around 60%, compared to an average placebo response rate of about 30%. Duloxetine has not been studied in the treatment of dysthymia, but has shown results in the treatment of major depression. In a 9-week, double-blind, placebo-controlled study of 257 patients with major depression, 65% responded to duloxetine 60mg/day, compared to 43% to placebo. Based on these results, it is highly likely that duloxetine will be an effective treatment for dysthymia.

This research study is being conducted at Stanford University Medical Center with a total of 24 patients, age 18 and above, with dysthymia.

In the study, subjects will receive duloxetine for 12 weeks. This is an open-label study, which means that every subject receives the study medication.

In total, subjects are seen for 10 visits across 13 weeks. At each visit subjects' heart rate, blood pressure and weight measurements will be obtained. At each visit study personnel will interview subjects about their symptoms, monitor side effects and ask them to complete study questionnaires.

Beginning at the second visit, subjects receive duloxetine 60 mg/day. If they experience side effects, the dose can be decreased to 30 mg/day for several days, but will be increased back to 60 mg/day by the end of the first week. If subjects are unable to tolerate a dose of 60 mg/day due to side effects, they will be withdrawn from the study. At the end of 6 weeks, if they have not responded to the study medication (as determined by doctor ratings based on subjects' reports), the dose of duloxetine will be increased to 120 mg/day, unless subjects are experiencing troubling side effects. Subjects continue on the minimum dose that brings about remission or the maximum tolerated dose for the remaining 6 weeks. Medication dosing will be flexible and determined by tolerance (side effects) and therapeutic effect.

ELIGIBILITY:
Inclusion Criteria::

* Sign an informed consent form
* 18 years of age or older
* Females not pregnant or breastfeeding or planning pregnancy and using an acceptable form of contraception
* Meet DSM-IV criteria for dysthymia
* A screening IDS-C score of 17 or greater
* No history of serious or unstable medical disorder
* Not taking any significant concurrent medications
* Not currently receiving psychotherapy Exclusion Criteria:- Suffering from DSM-IV defined
* delirium, dementia, amnestic, or other cognitive disorders
* mental disorders due to a general medical condition
* factitious or somatoform disorders
* mental retardation or developmental disabilities
* substance or alcohol abuse within the last 3 months
* depressive disorders with current suicidal risk
* psychotic disorders including delusional disorder, somatic type
* dissociative disorder
* personality disorders sufficiently severe to interfere with study participation
* History of DSM-IV defined bipolar I or II disorder
* History of non-response of dysthymia to adequate antidepressant medication
* History of major depression refractory to two adequate trials of antidepressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2004-09; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Inventory of Depressive Symptomatology (Clinician-Rated)

SECONDARY OUTCOMES:
Clinical Global Impressions - Improvement
Zung Self-Rating Depression Scale
Patient Global Improvement
Brief Pain Inventory
WHO-QOL 100

CONTACTS AND LOCATIONS:
Overall Officials: Lorrin M Koran, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Koran LM, Aboujaoude EN, Gamel NN. Duloxetine treatment of dysthymia and double depression: an open-label trial. J Clin Psychiatry. 2007 May;68(5):761-5. doi: 10.4088/jcp.v68n0514. PMID 17503986